CLINICAL TRIAL: NCT02575196
Title: Phase 2 Prospective, Observational, Pilot Study of Noninvasive Monitoring of Regional Cerebral Blood Flow for the Evaluation of Brain Tissue Perfusion During and After Resuscitation for Cardiac Arrest
Brief Title: Non Invasive Neuromonitoring After Cardiac Arrest
Acronym: NINCA
Status: Completed | Type: Observational
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Other Study IDs: GCO 15-1105
Record Dates: First submitted 2015-10-12; First posted 2015-10-14 (Estimated); Last update posted 2017-04-19 (Actual); Status verified 2017-04

CONDITIONS: Cardiac Arrest
Keywords: Cardiac arrest; Cardiopulmonary Resuscitation; CPR; cerebral blood flow; cerebral perfusion
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cardiac arrest: Consecutive adult cardiac arrest patients with sustained ROSC in an academic medical center
  Interventions: Device: Non-invasive cerebral flow monitoring

INTERVENTIONS:
Device: Non-invasive cerebral flow monitoring — As soon as possible after ROSC, c-flow monitor will be connected to the patient, recording cerebral flow index for the first 72 hours following ROSC. All other relevant clinical data will be recorded.
  Other Names: c-flow monitor (ORNIM)

SUMMARY:
Cardiac Arrest is among the leading causes of death, with survival still well under 50% and the majority of the survivors suffering from moderate to severe neurologic deficits. The human, social and economic costs are staggering.

During resuscitation, damage is mitigated if chest compressions and other medical care are optimal, allowing some blood to reach the brain and some oxygen to reach the cells. Once the heart starts beating again, which is called return of spontaneous circulation, brain perfusion is reestablished, but usually not to normal. The now damaged brain is very fragile, can be sensitive to any changes in blood pressure or metabolic abnormalities, and swelling might set in. Hypoperfusion can persist, without the clinician's knowledge. All of these events further damage the brain and diminish the odds that the patient will regain a normal life. Therefore, the hours following return to spontaneous circulation are critical to the patient's future recovery, and constitute a window of opportunity to maximize the brain ability to heal.

In order to optimize resuscitative efforts and post-arrest management, clinicians must know what is actually happening with the most vital organ, the brain. The problem is that it is very difficult to do in a comatose patient. The available technologies only reveal indirect evidence of brain suffering, like the swelling on CT-scans, but not to continuously evaluate at the bedside if the brain actually receives enough blood.

The FDA recently approved a device named the c-flow, made by ORNIM. This device looks at red blood cells in the brain and the speed at which they move to evaluate an index of cerebral perfusion. It does so with sensors put on the patient's forehead, which emit and detect ultrasounds and infrared light. This index can inform the clinician about the amount of blood flow the brain receives, and it can be put in place very quickly, even during resuscitative efforts, and without any danger for the patient.

The study looks at how well the information obtained with the c-flow matches the one obtained from other indirect indices and, more importantly, how well it predicts patient outcome. The investigators wish to establish threshold values of this index of perfusion that predict a good recovery so that this information may be used to optimize patient's neurological outcome in the near future.

DETAILED DESCRIPTION:
Primary Objective:

Cardio-Pulmonary Resuscitation (CPR) is undergoing a major paradigm shift, with new emphasis on optimizing neurological recovery. As a result, Cardio-Cerebral Resuscitation (CCR) is now the preferred term for describing protocols directed at promoting survival and recovery from cardiac arrest. Establishing and maintaining brain perfusion is the critical endpoint of resuscitation; however, there is currently no simple and reliable way to evaluate the adequacy of brain tissue perfusion in cardiac arrest patients. The overall goal of the NINCA study is to determine if non-invasive cerebral blood flow index (CFI) can be used as a simple and effective measurement of brain perfusion during and after resuscitation from cardiac arrest. Our researchers hypothesize that this monitoring may one day be routinely used to (1) evaluate the adequacy of chest compressions, (2) avoid brain tissue hypoperfusion induced by excessive hyperventilation or shivering, (3) serve as an endpoint for goal-directed hemodynamic support, (4) evaluate the potential for neurological recovery, and (5) help guide post-cardiac arrest care.

Implications for Further Research:

Successful completion of the research will hopefully establish that non- invasive cerebral blood flow monitoring is feasible during and after CPR; is dependent on adequate MAP, CO, temperature, SpO2 and ventilation; and is a valid predictor of neurological recovery. If confirmed, such monitors may one day become part of standard ICU post-cardiac arrest monitoring and even be part of standard resuscitation equipment.

Determination of optimal CFI thresholds or targets will support future studies to determine if "goal directed" and individualized post-resuscitation ICU care is feasible using non-invasive cerebral perfusion indices. This could lead to a new way of optimizing hemodynamic support, temperature management and ventilation strategies to maintain adequate cerebral perfusion and improve neurological outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Sustained ROSC within 60 minutes of arrest
* Patient is comatose (unresponsive and unable to follow verbal commands) after resuscitation

Exclusion Criteria:cerebral perfusion

* Partially or fully dependant functional status prior to index cardiac event
* Acute traumatic brain injury, SAH, massive stroke or intracranial hemorrhage
* Initiation of monitoring is not feasible for logistical reasons
* Urgent surgery planned
* Severe co-morbidity or terminal illness which makes survival to 3 months unlikely
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Comatose survivors of cardiac arrest
Sampling Method: Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2015-10; Primary Completion 2016-03-21 (Actual); Study Completion 2016-03-21 (Actual)

PRIMARY OUTCOMES:
Cerebral Performance Category | 7 days
  Neurological Outcome by good functional recovery
Modified Rankin Scale | 7 days
  Neurological Outcome

SECONDARY OUTCOMES:
Survival Rate | 7 days
  Survival with good functional recovery

OTHER OUTCOMES:
MoCA | 7 days
  Cognitive outcome
EQ-5L-5D | 7 days
  quality of life outcome

CONTACTS AND LOCATIONS:
Overall Officials: Stephan A Mayer, MD, Principal Investigator — Neurology Department, Mount Sinai Hospital
Locations (1):
- Mount Sinai Hospital, New York, New York, United States

REFERENCES:
- [Derived] Francoeur CL, Lee J, Dangayach N, Gidwani U, Mayer SA. Non-invasive cerebral perfusion monitoring in cardiac arrest patients: a prospective cohort study. Clin Neurol Neurosurg. 2020 Sep;196:105970. doi: 10.1016/j.clineuro.2020.105970. Epub 2020 May 30. PMID 32505869